CLINICAL TRIAL: NCT05146700
Title: Comparing Restrictive Vs. Liberal Oxygen Strategies for Trauma Patients: the TRAUMOX2 Trial
Brief Title: Restrictive Vs. Liberal Oxygen in Trauma
Acronym: TRAUMOX2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Jacob Steinmetz, MD, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6011; 2021-000556-19 (EudraCT Number); NNF20OC0063985 (Other Grant/Funding Number: Novo Nordisk Fonden)
Record Dates: First submitted 2021-11-30; First posted 2021-12-07 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Trauma; Oxygen Toxicity; Wounds and Injuries
Keywords: Trauma; Oxygen
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Trial participants are randomized pre-hospital or in the trauma bay to a restrictive or liberal oxygen treatment for eight hours.
  Experimental (restrictive oxygen): The restrictive group will receive the lowest dosage of oxygen (≥21%) ensuring an SpO2 target = 94%
  Active comparator (liberal oxygen): The liberal group will receive a flow of 15 L O2/min for non-intubated trial participants or an FiO2 = 1.0 for intubated trial participants in the pre-hospital phase, the trauma bay and during intrahospital transportation; later in the operating room (OR), intensive care unit (ICU), post-anesthesia care unit (PACU) and ward, the flow/FiO2 can be reduced to ≥12 L O2/min or FiO2 ≥0.6 if the arterial oxygen saturation (SpO2) is ≥98%
Who Masked: Outcomes Assessor
Masking Description: Open-label, primary outcome assessor- and analyst-blinded, randomized, controlled clinical trial with regards to treatment: treating staff will be aware of the trial participants' randomization group.
  While including patients for the study, the research team and treating staff will be aware of the trial participants' oxygen allocation strategy. However, at least two allocation blinded primary outcome assessors (specialists in anesthesiology, intensive care, emergency medicine or similar) will be appointed at each center to assess in-hospital major lung complications (pneumonia and acute respiratory distress syndrome). Blinding will be ensured by concealing all information indicative of the allocation prior to assessment. The statistician and manuscript writers will be blinded towards the allocation of treatment once the trial ends when data is being analysed and the manuscript is drafted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive oxygen (Experimental): - Lowest oxygen delivery possible (≥21%) ensuring an SpO2 target = 94% either using no supplemental oxygen, a nasal cannula, a non-rebreather mask or manual/mechanical ventilation (intubated trial participants)
  and
  - Only trial participants receiving an FiO2 = 0.21 can saturate >94%
  Pre-oxygenation as usual prior to intubation is permitted
  Interventions: Drug: Restrictive oxygen
- Liberal oxygen (Active Comparator): - 15 L O2/min flow for non-intubated trial participants in the pre-hospital phase, the trauma bay and during intrahospital transportation. In the operating room, intensive care unit, post-anesthesia care unit and ward the flow can be reduced to ≥12 L O2/min if the arterial oxygen saturation is ≥98%
  or
  - FiO2 = 1.0 for intubated trial participants in the pre-hospital phase, the trauma bay and during intrahospital transportation. In the operating room, intensive care unit, post-anesthesia care unit and ward the FiO2 can be reduced to ≥0.6 if the arterial oxygen saturation is ≥98%
  Interventions: Drug: Liberal oxygen

INTERVENTIONS:
Drug: Restrictive oxygen — Lowest oxygen delivery possible (≥21%) ensuring an SpO2 target = 94%
  Arms: Restrictive oxygen
Drug: Liberal oxygen — 15 L O2/min flow for non-intubated trial participants or FiO2 = 1.0 for intubated trial participants in the initial phase; later in the operating room, intensive care unit, post-anesthesia care unit and ward, the flow/FiO2 can be reduced to ≥12 L O2/min or FiO2 ≥0.6 if the arterial oxygen saturation is ≥98%
  Arms: Liberal oxygen

SUMMARY:
Victims of trauma are often healthy individuals prior to the incident, but acquire numerous complications including sepsis and pulmonary complications and diminished quality of life after trauma. According to Advanced Trauma Life Support guidelines, all severely injured trauma patients should receive supplemental oxygen.

The objective of TRAUMOX2 is to compare the effect of a restrictive versus liberal oxygen strategy the first eight hours following trauma on the incidence of 30-day mortality and/or major respiratory complications (pneumonia and acute respiratory distress syndrome) within 30 days (combined primary endpoint).

DETAILED DESCRIPTION:
In trauma resuscitation, supplemental oxygen is often administered both to treat and prevent hypoxemia as recommended both by the Advanced Trauma Life Support (ATLS) manual and the Pre-hospital Trauma Life Support (PHTLS) manual. Oxygen is administered in many other situations too, sometimes in a non-consistent manner and very often without even being prescribed. In a recent systematic review, our group found the evidence both for and against the use of supplemental oxygen in the trauma population to be extremely sparse. However, a recent systematic review and meta-analysis comparing liberal versus restrictive oxygen strategy for a broad mix of acutely ill medical and surgical patients found an association between liberal oxygen administration and increased mortality. Of note, only one small study on trauma patients (patients with traumatic brain injury), which did not report mortality data, was included. Conversely, this study showed that degree of disability was significantly reduced at six months in the group receiving liberal compared to restrictive oxygen.

In mechanically ventilated patients hyperoxemia is commonly observed (16-50%), and hyperoxemia is a common finding in trauma patients in general. In addition to mortality, hyperoxemia has been associated with major pulmonary complications in the Intensive Care Unit (ICU) as well as in surgical patients. For example, a recent retrospective study found hyperoxemia to be an independent risk factor for ventilator associated pneumonia (VAP). Nevertheless, a highly debated recommendation from the World Health Organisation strongly recommends that adult patients undergoing general anesthesia for surgical procedures receive a fraction of inspired oxygen (FiO2) of 80% intraoperatively as well as in the immediate postoperative period for two to six hours to reduce the risk of surgical site infection. Furthermore, a study on 152,000 mechanically ventilated patients found no association between hyperoxia and mortality during the first 24 hours in the ICU, and another study on 14,000 mixed ICU patients found that a partial arterial oxygen pressure (PaO2) of approximately 18 kPa resulted in the lowest mortality. Finally, a recent study randomized 2928 ICU patients to either low or high oxygenation (defined as 8 vs 12 kPa) for a maximum of 90 days and found no difference in mortality. Therefore, whether the trauma population could benefit from a more restrictive supplemental oxygen approach than recommended by current international guidelines presents a large and important knowledge gap.

In a recent pilot randomized clinical trial (TRAUMOX1, ClinicalTrials.gov Registration number: NCT03491644), we compared a restrictive and a liberal oxygen strategy for 24 hours after trauma (N = 41) and found maintenance of normoxemia following trauma using a restrictive oxygen strategy to be feasible. TRAUMOX1 served as the basis for this larger trial. We experienced 24 hours to be slightly excessive to represent only the acute phase post trauma for which reason we have shortened the time-period to eight hours in TRAUMOX2. Furthermore, we found that several physicians had important concerns with the high dosage of oxygen in the liberal arm for which reason the concentration will be reduced. Finally, we did not randomize trauma patients in the pre-hospital phase, but instead on arrival at the trauma bay (median [interquartile range (IQR)] time to randomization: 7 [4-10] minutes, median [IQR] time from trauma to trauma bay arrival: 51 [29.0-67.5] minutes). To limit this inconsistent exposure to oxygen in the pre-hospital phase prior to inclusion we will initiate the intervention in the pre-hospital phase where possible in TRAUMOX2.

The objective of TRAUMOX2 is to compare the effect of a restrictive versus liberal oxygen strategy the first eight hours following trauma on the incidence of 30-day mortality and/or major respiratory complications (pneumonia and acute respiratory distress syndrome) within 30 days (combined primary endpoint).

We hypothesize that a restrictive compared to a liberal oxygen strategy for the initial eight hours after trauma will result in a lower rate of 30-day mortality and/or major respiratory complications (pneumonia and acute respiratory distress syndrome) within 30 days (combined primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years, including fertile women
* Blunt or penetrating trauma mechanism
* Direct transfer from the scene of accident to one of the participating trauma centers
* Trauma team activation
* The enrolling physician must initially expect a hospital length of stay for 24 hours or longer

Exclusion Criteria:

* Patients in cardiac arrest before or on admission
* Patients with a suspicion of carbon monoxide intoxication
* Patients with no/minor injuries after secondary survey will be excluded if they are expected to be discharged <24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1508 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-10-12 (Actual)

PRIMARY OUTCOMES:
The incidence of 30-day mortality and/or major respiratory complications (pneumonia and acute respiratory distress syndrome) within 30 days (combined primary endpoint) | Day 30 after enrollment
  The assessment of the major respiratory complications will be performed by at least two allocation blinded primary outcome assessors (specialists in anesthesiology, intensive care, emergency medicine or similar); blinding will be ensured by concealing all information indicative of the allocation prior to assessment

SECONDARY OUTCOMES:
30-day mortality | Day 30 after enrollment
  Assessed in the patient's medical record/register
12-month mortality | 12 months after enrollment
  Assessed in the patient's medical record/register
Major respiratory complications (pneumonia and acute respiratory distress syndrome) within 30 days | Day 30 after enrollment
  Data from the combined primary endpoint assessment
Hospital length of stay | From date of admission to discharge from the hospital, up to 12 months after enrollment
  Number of days
ICU length of stay | From date of admission to discharge from the ICU, up to 12 months after enrollment
  Number of days
Time on mechanical ventilation | From initiation of mechanical ventilation to being ventilator-free within 30 days after enrollment
  Number of hours; only mechanical ventilation in the ICU should be considered
Days alive outside the ICU | ICU-free days within 30 days after enrollment
  Number of days
Days alive without mechanical ventilation | Ventilator-free days within 30 days after enrollment
  Number of days; only mechanical ventilation in the ICU should be considered
Re-intubations | Within 30 days after enrollment
  Number of re-intubations; only re-intubations in the ICU should be considered
Pneumonia post-discharge | From discharge to a maximum of 30 days after enrollment
  Number of trial participants; evaluated through medicines prescribed after hospital discharge in countries where this information is available
Episode(s) of hypoxemia during intervention (saturation <90%) | During the 8 hours of the oxygen intervention arms
  Defined as number of times the valid oxygen saturation is below 90%; if it is below 90%, above 90% and below 90% again, then it should be registered as 2 episodes
Surgical site infections | Within 30 days after enrollment
  Defined as per the Centers for Disease Control and Prevention (CDC) criteria for a surgical site infection event
5-level EQ-5D version (EQ-5D-5L) score | 6 and 12 months post-trauma
  Conducted through a telephone interview where the patient is asked to indicate his/her health state
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS)
  The EQ-5D descriptive system consists of a scale (minimum score = 5 and maximum score = 25) where the lowest score (5) indicates no problems whereas the highest score (25) indicates extreme problems
  The EQ VAS (visual analogue scale) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled "The worst health you can imagine" (minimum score = 0) and "The best health you can imagine' (maximum score = 100)
The Glasgow Outcome Scale Extended (GOSE) score | 6 and 12 months post-trauma
  Conducted through a telephone interview where the patient/patient's next-of-kin/caretaker is interviewed through a structured questionnaire to assess the functional recovery after trauma
  The GOSE consists of a scale (minimum value = 1 and maximum value = 8); each patient given a score based on the interview:
  1 = Death, 2 = Vegetative state, 3 = Lower severe disability, 4 = Upper severe disability, 5 = Lower moderate disability, 6 = Upper moderate disability, 7 = Lower good recovery, 8 = Upper good recovery
Levels of oxidative stress biomarkers, primarily malondialdehyde (MDA) at hour 24 | Hour 0, hour 8, hour 24 and hour 48 after enrollment
  The unit of the oxidative stress biomarker depends on the chosen analysis of the specific biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Steinmetz, MD, PhD, Study Director — Consultant; Tobias Arleth, MD, Principal Investigator — Research assistent
Locations (5):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense
- Erasmus MC, University Medical Center Rotterdam, Rotterdam, Rotterdam, Netherlands
- Inselspital University Hospital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Arleth T, Baekgaard J, Siersma V, Creutzburg A, Dinesen F, Rosenkrantz O, Heiberg J, Isbye D, Mikkelsen S, Hansen PM, Zwisler ST, Darling S, Petersen LB, Morkeberg MCR, Andersen M, Fenger-Eriksen C, Bach PT, Van Vledder MG, Van Lieshout EMM, Ottenhof NA, Maissan IM, Den Hartog D, Hautz WE, Jakob DA, Iten M, Haenggi M, Albrecht R, Hinkelbein J, Klimek M, Rasmussen LS, Steinmetz J; TRAUMOX2 Trial Group. Early Restrictive vs Liberal Oxygen for Trauma Patients: The TRAUMOX2 Randomized Clinical Trial. JAMA. 2025 Feb 11;333(6):479-489. doi: 10.1001/jama.2024.25786. PMID 39657224
- [Derived] Arleth T, Baekgaard J, Siersma V, Klimek M, Hinkelbein J, Rasmussen LS, Steinmetz J; TRAUMOX2 Study Group. Comparing restrictive versus liberal oxygen strategies for trauma patients: The TRAUMOX2 trial-Statistical analysis plan. Acta Anaesthesiol Scand. 2023 Jul;67(6):829-838. doi: 10.1111/aas.14230. Epub 2023 Mar 28. PMID 36906804
- [Derived] Baekgaard J, Arleth T, Siersma V, Hinkelbein J, Yucetepe S, Klimek M, van Vledder MG, Van Lieshout EMM, Mikkelsen S, Zwisler ST, Andersen M, Fenger-Eriksen C, Isbye DL, Rasmussen LS, Steinmetz J. Comparing restrictive versus liberal oxygen strategies for trauma patients - the TRAUMOX2 trial: protocol for a randomised clinical trial. BMJ Open. 2022 Nov 7;12(11):e064047. doi: 10.1136/bmjopen-2022-064047. PMID 36344005
- See also: The official study website of TRAUMOX2 — https://www.traumox2.org